CLINICAL TRIAL: NCT01663025
Title: Evaluating The Effects Of Intra Operative Hand Reflexology on Pain and Anxiety During Out Patient Vein Surgery
Brief Title: The Effects of Intra Operative Hand Reflexology for Patients Receiving Out Patient Vein Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WC1HM
Record Dates: First submitted 2012-08-06; First posted 2012-08-13 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Anxiety
Keywords: Randomised controlled trial; Pain; Anxiety; Ambulatory surgery; Hand massage; Local anaesthetic
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hand Reflexology (Experimental): Participants in this condition will receive hand reflexology, performed by a trained reflexologist during their treatment. This will be in addition to usual standard care therefore the surgeon will speak to the participant occasionally to ensure they are comfortable.
  Interventions: Behavioral: Hand Reflexology
- Control (No Intervention): Participants in condition will form the control group for the study. They will receive usual standard care during treatment which will involve the surgeon speaking to them occasionally to ensure that they are comfortable.

INTERVENTIONS:
Behavioral: Hand Reflexology — The hand reflexology will begin in theatre, before the local anaesthetic is administered and will continue until the patient is ready to leave the operating theatre.
  Arms: Hand Reflexology

SUMMARY:
This randomised controlled trial aims to compare the effectiveness of hand reflexology received during office based vein surgery, under local anaesthetic on patient's reports of pain and anxiety, compared to usual standard care.

DETAILED DESCRIPTION:
The negative effects of anxiety and pain on surgical recovery are well documented. It is also accepted that distraction can be effective in pain reduction. This randomised controlled trial will explore the effect of intra operative hand reflexology on pain perception and anxiety during office-based surgery under local anaesthetic. Participants will be randomly allocated to either the experimental condition, in which they will receive a hand reflexology during treatment, or control condition in which they will receive usual standard care. Immediate and longer term outcomes will be explored.

Eight weeks after surgery, participants will return to the clinic for a follow up appointment. While they are in the waiting area they will be asked to complete a short questionnaire to assess time taken to return to pre surgical levels of functioning, pain experienced in the first four weeks after surgery, severity of venous symptoms and satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* To be aged between 18 and 80
* To be able to give informed consent
* To be receiving, endovenous laser ablation or phlebectomies for the treatment of varicose veins
* To have a good understanding of written and spoken English.
* To arrive at the clinic with sufficient time before their procedure to give consent and complete the questionnaire (>20 mins)

Exclusion Criteria:

-To be aged under 18 or over 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pain | In the recovery area, immediately after surgery
  Participants will complete a numeric rating scale (0 no pain - 10, extreme pain) to assess any painful sensations experienced during treatment

SECONDARY OUTCOMES:
Anxiety | In the recovery area, immediately after surgery
  Participants will complete a numeric rating scale(0, no anxiety to 10, extreme anxiety)to assess any anxiety they experienced during treatment.
Satisfaction with treatment | in the recovery area, immediately after surgery
  Participants will be asked to rate how satisfied they are with the treatment that they have received on a scale of 1 (very dissatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Whiteley, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic at the Wimpole Clinic, London, London, United Kingdom